CLINICAL TRIAL: NCT01100151
Title: A Phase 2 Study of the Effects of RDC-1036 Administered to Subjects With Opioid-induced Constipation During Treatment With Opioids for Chronic Pain
Brief Title: ALK37-003: A Study of RDC-1036 (ALKS 37) in Adults With Opioid-induced Constipation (OIC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK37-003
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Opioid-induced Constipation
Keywords: Opioid-induced constipation; RDC-1036; ALKS 37
MeSH Terms: conditions — Opioid-Induced Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RDC-1036 (ALKS 37) (Experimental): Capsules for oral administration
  Interventions: Drug: RDC-1036 (ALKS 37)
- Placebo (Placebo Comparator): Capsules for oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RDC-1036 (ALKS 37) — Capsules for oral administration
  Arms: RDC-1036 (ALKS 37)
Drug: Placebo — Capsules for oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of RDC-1036 (ALKS 37) in adults with opioid-induced constipation (OIC) following repeat dose administration

DETAILED DESCRIPTION:
Approximately 60 subjects will be enrolled in 1 of 2 cohorts. Following a review of Cohort 1 safety and tolerability data, subjects will then be enrolled into Cohort 2, to explore additional doses. Dose escalation will occur in both cohorts. There will be 18 visits over a 6-week period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Body mass index (BMI) of 19 to 35 kg/m2 at screening
* Receiving prescribed opioid medication for the management of chronic, non-cancer, pain
* Diagnosis of opioid-induced constipation (OIC)
* Willingness to stop all laxatives and other bowel regimens from the first study visit following screening until the end of the study. The use of constipation rescue medication will be allowed during the study.

Exclusion Criteria:

* Pregnancy and/or currently breastfeeding
* Clinically significant medical condition or illness (other than the condition for which the pain medication is being prescribed)
* Receiving treatment with opioid therapy for cancer-related pain, abdominal pain, scleroderma, and/or for the management of drug addiction
* Any gastrointestinal (GI) or pelvic disorder known to affect bowel transit, produce a GI obstruction, or contribute to bowel dysfunction other than opioid-induced constipation (eg, diverticulitis, other intestinal strictures, bezoars)
* Use of medical devices such as pacemakers, infusion pumps, or insulin pumps
* Use of naloxone, Subutex or Suboxone, Revia, Relistor, or Entereg starting 15 days before the first study visit following screening until the end of the study
* Participation in a clinical trial of a pharmacological agent within 30 days before screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in frequency of spontaneous bowel movement (SBM) from pre-treatment period to treatment period | 4 Weeks
Number of subjects reporting treatment-emergent adverse events (TEAEs) | 6 Weeks
  A TEAE is any adverse event (AE), whether or not considered drug-related, that develops or worsens in severity after study drug administration begins (ie, from the first administration through the end of the follow-up period).

SECONDARY OUTCOMES:
Change in rescue laxative use from pre-treatment to treatment period | 4 Weeks
Study drug dose prior to first SBM after randomization | 4 weeks
Scores to study-related questionnaires | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.
Locations (11):
- United States (11):
  - Alkermes Investigational Site, Sheffield, Alabama
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Pasadena, California
  - Alkermes Investigational Site, Walnut Creek, California
  - Alkermes Investigational Site, DeLand, Florida
  - Alkermes Investigative Site, New Smyrna Beach, Florida
  - Alkermes Investigational Site, Boise, Idaho
  - Alkermes Investigational Site, New Orleans, Louisiana
  - Alkermes Investigational Site, Winston-Salem, North Carolina
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Salt Lake City, Utah